CLINICAL TRIAL: NCT03967483
Title: Non Interventional Study on Indomethacin-responsive Headaches
Brief Title: Study on Indomethacin-responsive Headaches
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anne Ducros (Other)
Responsible Party: Sponsor-Investigator, Anne Ducros, Pr, French Society for the Study of Migraine Headache
Organization: French Society for the Study of Migraine Headache (Other)
Other Study IDs: 2019-A00406-51
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Indomethacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Indometacin — patient who are taken indomatacin for headaches and migraine

SUMMARY:
Description of modalities concerning the patient care of headaches sensible to indometacine.

DETAILED DESCRIPTION:
Description of clinical profile, treatment of crisis and background treatment

ELIGIBILITY:
Inclusion Criteria:

* patient with a diagnosis of migraine with or without aura, or trigemino-autosomic headaches or other primary headaches
* patient who are taking indometacine
* patient with written consent form

Exclusion Criteria:

* patient under 18 years
* pregnant woman or breastfeeding patient
* patient who refuses to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient sufffuring from headaches or migraine and who is receiving Indometacine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Description of headaches sensible to indometacine | 24 monthes
  Description of the clinical cases with headaches sensible to indometacine according to the type of headaches.